CLINICAL TRIAL: NCT04618965
Title: The Effect of Intrathecal Versus Intravenous Dexmeditomedine on Postoperative Analgesia in Transurethral Resection of the Prostate
Brief Title: Intrathecal Versus Intravenous Dexmeditomedine in Transurethral Resection of the Prostate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Laila Elahwal, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pain relief for prostatictomy
Record Dates: First submitted 2020-10-26; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Dexmedetomidine; Transurethral Resection of Prostate; Intravenous; Intrathecal
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo) group (Placebo Comparator): Each patient will receive intrathecal hyperbaric bupivacaine 10 mg in 2.5 ml and 0.5 ml saline with 3 mL total volume. Continous 50 ml saline infusion for 10 min followed by 200 ml saline infusion till the end of surgery.
  Interventions: Drug: control group
- Intrathecal dexmedetomidine group (Experimental): Each patient will receive dexmedetomidine 5 μg diluted in 0.5ml saline and hyperbaric Bupivacaine 10 mg in 2.5 ml with 3 mL total volume. Continous 50 ml saline infusion for 10 min followed by 200 ml saline infusion till the end of surgery.
  Interventions: Drug: Intrathecal dexmedetomidine
- Intravenous dexmedetomidine group (Experimental): Each patient will receive intravenous dexmedetomidine started at a loading dose of 1 μg/kg diluted in 50 ml saline and administered within 10 min as a loading dose, followed by maintenance at a dose of 0.4 μg/kg/h diluted in 200 ml saline till the end of surgery and hyperbaric Bupivacaine 10 mg in 2.5 ml total volume.
  Interventions: Drug: Intravenous dexmedetomidine

INTERVENTIONS:
Drug: control group — Each patient will receive intrathecal hyperbaric bupivacaine 10 mg in 2.5 ml and 0.5 ml saline with 3 mL total volume. Continous 50 ml saline infusion for 10 min followed by 200 ml saline infusion till the end of surgery.
  Arms: Control (Placebo) group
Drug: Intrathecal dexmedetomidine — Each patient will receive dexmedetomidine 5 μg diluted in 0.5ml saline and hyperbaric Bupivacaine 10 mg in 2.5 ml with 3 mL total volume. Continous 50 ml saline infusion for 10 min followed by 200 ml saline infusion till the end of surgery.
  Arms: Intrathecal dexmedetomidine group
Drug: Intravenous dexmedetomidine — Each patient will receive intravenous dexmedetomidine started at a loading dose of 1 μg/kg diluted in 50 ml saline and administered within 10 min as a loading dose, followed by maintenance at a dose of 0.4 μg/kg/h diluted in 200 ml saline till the end of surgery and hyperbaric Bupivacaine 10 mg in 2.5 ml total volume.
  Arms: Intravenous dexmedetomidine group

SUMMARY:
This study is to evaluate The analgesic effect of intrathecal versus intravenous dexmeditomedine in transurethral resection of the prostate

DETAILED DESCRIPTION:
This study will carried out in Tanta University hospital on75 male patients Patients will randomly classified into 3 groups Group I: will receive intrathecal hyperbaric bupivacaine 10mg in 2.5 ml and .5 ml saline with 3ml total volume Group II: will receive dexmeditomedine 5Mic diluted in.5 ml saline and hyperbaric bupivacaine 10mg in 2.5ml with 3ml total volume Group IIl: Will receive intravenous dexmeditomedine started at loading dose of 1 mic/kg diluted in 50 ml saline and administered within 10 min as loading dose , followed by maintenance at a dose of .4mic/kg/h diluted in200 ml saline till the end of surgery and hyperbaric bupivacaine 10 mg in 2.5 ml total volume

ELIGIBILITY:
Inclusion Criteria:

* male gender
* 50:70years old
* ASA:I,II

Exclusion Criteria:

* contraindications of spinal anesthesia
* Patient refusal
* Patient taking alpha agonist or antagonist
* Uncontrolled cardiac diseases
* Allergy to local anesthetic drugs

Ages: 59 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-04-26 (Estimated); Study Completion 2021-06-26 (Estimated)

PRIMARY OUTCOMES:
The time to first rescue analgesic | 24 hours postoperative
  The duration between the administration of spinal block and the first desire for supplemental analgesia (onset of 1st post-operative analgesic dose).
  First post-operative analgesic dose will be1 μg/kg intravenous fentanyl when visual analogue pain score (VAS) is 4 or more

SECONDARY OUTCOMES:
Postoperative pain score Total dose of analgesic consumption I the first postoperative day Intraoperative and postoperative complications | 24 hours postoperative
  Visual analogue score (VAS) between 0 and 10{0= no pain, 10=most severe pain}
Total analgesic consumption | 24 hours postoperative
  The pain score will be assessed every 4 h in 24 h and fentanyl will be given in a dose of 1 μg /kg when Visual analogue score (VAS) is 4 or more. Any out breaking pain will be treated with increments of fentanyl in a dose of 0.5μg/kg.
Intraoperative and postoperative complications | Intraoperative and 24 hours postoperative
  e.g. hypotension, bradycardia and vomiting

IPD SHARING:
Plan to Share IPD: No